

# **CONFIDENTIAL - PROTOCOL**

The following contains confidential, proprietary information which is the property of Recros Medica

The PREFORM Study: An Exploratory, Single-Center Study to Evaluate the Safety and Efficacy of Rotational Fractional Resection on Submental Contouring and Optimal Peri-Procedure Regimen for Accelerated Recovery

Protocol Number: CLP-0007

Version 17-May-2019, Amendment 1

Name of Investigational Product: Recros Medica Focal Contouring System

Sponsor: Recros Medica, Inc.

3525 Del Mar Heights Road, Suite 609

San Diego, CA 92130a

Emergency Telephone Number(s): 714-309-7667

Serious Adverse Event Reporting: rmcintosh@recrosmedica.com

Recros Medica Safety Physician: Catherine Kusnick, MD

Recros Medica Signatory: Robin McIntosh

NCT Number: NCT03966924

#### **Investigational Device:**

Recros Medica Focal Contouring System to perform Rotational Fractional Resection (skin resection with and without and focal lipectomy)

#### **Study Objective:**

The objective is to explore and evaluate the peri-procedure treatment plan for accelerated recovery after Rotational Fractional Resection in patients with submental laxity.

### **Study Design**

*Structure*: Prospective, single-center, exploratory, interventional cohort, non-significant risk (NSR) study.

Duration: Approximately 4 months for each subject from the screening visit to the exit visit.

*Visit Schedule*: Screening, procedure, Day 1, 4, 7, 14, 21, 30, 45, 60, and 90 post-procedure. An optional visit may occur 5-6 days after procedure.

*Indication for Use*: The Recros Medica focal contouring system is intended for resecting skin with and without fat removal for the purpose of submental contouring.

## **Study Population Characteristics**

*Number of Subjects*: Up to approximately 50 subjects will be enrolled (consented) to ensure up to approximately 30 subjects treated at 1 US site.

Condition/Disease: Adult subjects with moderate to severe submental laxity.

Key Inclusion Criteria: Healthy male or female, at least 30 years old; moderate to severe submental laxity; agree to maintain weight  $(\pm 5\%)$  for the duration of the study

Key Exclusion Criteria: History of psoriasis, hyperpigmentation, eczema, rosacea or vitiligo; history of keloids, hypertrophic scarring, or other skin condition that may result in excessive scarring; Fitzpatrick skin type 4, 5, and 6; severe or very severe lipodystrophy; body mass index >30 kg/m²; treatment with aspirin or aspirin containing products (e.g., Excedrin), NSAIDS, vitamin E within 14 days of the procedure.

#### **Response Measures**

## Efficacy:

- Submental Skin Laxity Scale, as assessed by the investigator
- Submental Lipodystrophy Scale, as assessed by the investigator
- Subject Satisfaction Questionnaire, as assessed by the subjects

## Safety:

- Visual Skin Assessment in the procedure area, as assessed by the investigator
- Visual Skin Assessment in procedure area by the subject
- Adverse events
- Manchester Scar Scale
- Visible scarring
- Pain assessment, using an 11-point Numeric Rating Scale (0 to 10), as assessed by the subject
- Vital signs (blood pressure and pulse rate)

#### Other:

- Peri-procedure interventions
- Elastic Adhesive Membrane Questionnaire
- Weight
- Photography

#### **Sample Size Calculation and Analysis Methods:**

Because this study is exploratory in nature, no sample size estimates have been performed.